CLINICAL TRIAL: NCT05652361
Title: Machine Learning-based Surgical Guidance System for Robot-assisted Rectal Surgery - a First-in-human Interventional Study
Brief Title: Machine Learning-based Surgical Guidance System for Robot-assisted Rectal Surgery
Acronym: CoBot2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Technische Universität Dresden (Other)
Collaborators: German Cancer Research Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TUD-COBOT2-087; DE-25-00015527 (Other: DMIDS)
Record Dates: First submitted 2022-12-07; First posted 2022-12-15 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Rectum Cancer
Keywords: Robotic Surgery; Total mesorectal excision
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Additional visualisation of surgical assistance during surgery (Experimental)
  Interventions: Other: Additional visualisation of surgical assistance during surgery

INTERVENTIONS:
Other: Additional visualisation of surgical assistance during surgery — Robot-assisted anterior rectal resection using daVinci® system as CE-marked gold standard with additional visualization of surgical assistance functions based on machine learning techniques

SUMMARY:
The aim of the study is to evaluate the technical feasibility and applicability of a surgical assistance system based on image recognition algorithms in a first-in-human pilot study. In addition, this study will provide preliminary data on the oncological outcome of the assistance system.

ELIGIBILITY:
Inclusion Criteria:

* Patients with rectal cancer scheduled for robot-assisted rectal resection
* Intact preoperative urogenital/rectal function
* Full capability of consent

Exclusion Criteria:

* Previous/Second malignant disease <5 years before diagnosis of rectal cancer
* Previous abdominal surgery, except for laparoscopic appendectomy, laparoscopic cholecystectomy or Cesarean section
* Pregnant or breastfeeding women
* Addiction or illness that prevent the person concerned from assessing the nature and scope of the clinical trial and its possible consequences
* indication that the participant is unlikely to comply with the trial protocoll (e.g. lack of compliance)
* official or court order for involuntary hospitalization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of discrepancies between the surgeon's preparation and the prediction of the CoBot system | 72 hours after Surgery
  System discrepancy score quantifying major misspecifications of the CoBot system in comparison to the surgeon's action

SECONDARY OUTCOMES:
Operating time [min] | During Surgery
  Time from skin incision until placement of last skin staple/suture
Duration of postoperative hospital stay [days] | At day of discharge, assessed up to 5 days
  Postoperative day 1 until day of discharge
Duration of postoperative intermediate/intensive care unit stay [days] | At day of discharge, assessed up to 5 days
  Postoperative day 1 until day of discharge
Frequency of peri-operative morbidity after resection | At day of discharge, assessed of up to 5 days
  Frequency of peri-operative complications after surgery until Day of Discharge
Kind of peri-operative morbidity after resection | At day of discharge, assessed of up to 5 days
  Kind of peri-operative complications after surgery until day of discharge
Assessment of the circumferential resection margin (CRM) | At day of discharge, assessed up to 5 days
  Rate of R0 resections
Number of resected lymphnodes | During surgery
  Number of lymphnodes resected during surgery
Assessment of pelvic function before and after rectal resection | 15 months
  Rectal function will be assessed preoperatively and 12-15 months postoperatively using the standard LARS score questionnaire, resulting in a score between 0 and 42. Higher scores mean a worse outcome (worse pelvic function).
Rectal sphincter function before and after rectal resection | 15 months
  Sphincter function will be assessed by manometry preoperatively and 12 - 15 months postoperatively
Assessment of the difficulty of the preparation | 48 hours after surgery
  Surgeon questionnaire, the questionnaire qualitatively assesses nine items, each item scoring from "not at all" to "very much", evaluated individually
Assessment of usability of guidance system | Through study completion, an average of 6 months
  One-time final survey of all participating surgeons, the questionnaire qualitatively assesses nine items, each item scoring from "not at all" to "very much", evaluated individually

CONTACTS AND LOCATIONS:
Overall Officials: Marius Distler, Prof. Dr., Principal Investigator — University Hospital Carl Gustav Carus Dresden
Locations (1):
- Department of Visceral, Thoracic and Vascular Surgery University Hospital Carl Gustav Carus Technische Universität Dresden, Dresden, Saxony, Germany

IPD SHARING:
Plan to Share IPD: No